CLINICAL TRIAL: NCT06622902
Title: Influence of Flow Rate Change on CO2 Levels During High Flow Nasal Ventilation (HFNV) in Preterm Infants.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Ori Hochwald , MD, Head, NICU, Rambam Health Care Campus
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RMB059422
Record Dates: First submitted 2024-06-26; First posted 2024-10-02 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Distress Syndrome; Prematurity; Non Invasive Ventilation
Keywords: Respiratory distress syndrome; prematurity; HIGH FLOW; CO2; VENTILATION
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- start with 2LPM (Experimental): start with 2LPM
  Interventions: Other: change flow from 6 to 2 LPM. Follow TcCO2 for 3 hours; Other: change flow from 2 to 6 LPM. Follow TcCO2 for 3h
- start with 6LPM0 (Experimental): start with 6LPM
  Interventions: Other: change flow from 6 to 2 LPM. Follow TcCO2 for 3 hours; Other: change flow from 2 to 6 LPM. Follow TcCO2 for 3h

INTERVENTIONS:
Other: change flow from 6 to 2 LPM. Follow TcCO2 for 3 hours — change flow from 6 to 2 LPM. Follow TcCO2 for 3 hours
Other: change flow from 2 to 6 LPM. Follow TcCO2 for 3h — change flow from 2 to 6 LPM. Follow TcCO2 for 3h

SUMMARY:
Background Preterm infants often need respiratory support. HFNV is a non-invasive method with benefits over CPAP, such as reduced nasal trauma and improved feeding.

Aim Study the impact of low (2 LPM) vs. high (6 LPM) HFNV flow rates on CO2 levels in preterm infants.

Methods Design: Prospective, crossover observational study. Participants: Preterm newborns (24-33.6 weeks' gestation) on HFNV. Procedure: Randomized flow rate adjustments, monitoring tcCO2 and other respiratory parameters over three hours.

Outcomes Primary: Change in tcCO2. Secondary: Study terminations due to unsafe CO2 levels and changes in other respiratory metrics.

Statistical Analysis Sample size: 45 infants. Analysis: Paired and unpaired t-tests for comparison within and between groups.

DETAILED DESCRIPTION:
Background:

Preterm Births: About 10% of births are preterm, with infants at risk for respiratory distress.

Respiratory Support: Endotracheal ventilation has improved survival but increased the risk of bronchopulmonary dysplasia.

Non-Invasive Support: Nasal CPAP minimizes complications. Heated, humidified high-flow nasal ventilation (HFNV) is an alternative, providing advantages like reduced nasal trauma and improved oral feeding.

Aim:

Primary Goal: Examine changes in transcutaneous CO2 (tcCO2) levels in preterm infants when using HFNV at low (2 LPM) versus high (6 LPM) flow rates.

Hypothesis: Different HFNV flow rates will show minimal change in tcCO2 (≤5 mmHg).

Methods:

Design: Prospective, crossover observational study in Rambam NICU. Participants: Preterm newborns (24-33.6 weeks' gestation) needing HFNV. Inclusion Criteria: Stabilized HFNP settings and tcCO2, parental consent. Exclusion Criteria: Specific flow and CO2 levels, unstable conditions, or congenital malformations.

Procedure: Randomize infants into two groups starting with 2 or 6 LPM flow rates, monitoring tcCO2 over three consecutive hours with alternating flow rates.

Measurements:

Primary Outcome: Change in tcCO2 levels. Secondary Outcomes: Number of study terminations due to pCO2/TcCO2 out of safety range, changes in respiratory parameters, and episodes of desaturation or bradycardia.

Statistical Analysis:

Sample Size: 45 infants needed to detect no difference with 90% power and 5% significance level.

Data Analysis: Use paired and unpaired Student's t-tests to compare results within and between groups.

Safety Protocol: The study will terminate if significant desaturation, bradycardia, or pCO2 levels outside the safety range occur.

ELIGIBILITY:
Inclusion criteria:

* Gestational age 240 to 336.
* At least 6 hours of stabilized HFNP settings, i.e. minor changes in settings (FiO2 ≤0.10, no change in flow).
* At least 6 hours of stabilized tcCO2, i.e. ≤5 mmHg variation.
* At least 6 hours from surfactant administration.
* Parental consent

Exclusion criteria:

* If flow is <3 and tcCO2 related pCO2 is<40mmHg.
* If Flow is ≥5 bpm and tcCO2 related pCO2 is>60mmHg.
* Unstable infants due to acute conditions (sepsis. IVH), or congenital malformations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Delta CO2 | 3 hours after flow change
  the change in TcCO2

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided